CLINICAL TRIAL: NCT01907672
Title: The Role of Rapid Diagnostic Tests for Malaria for Targeting of ACTs at Community Level: a Cluster Randomized Trial
Brief Title: The Role of Rapid Diagnostic Tests for Malaria for Targeting of ACTs at Community Level
Acronym: GhanaCommRDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ghana Health Services (Other Government)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Evelyn K. Ansah, Deputy Director (Research), Ghana Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ITDCVT68; MCDC_SF_02 (Other Grant/Funding Number: Malaria Capacity Development Consortium (MCDC))
Record Dates: First submitted 2012-09-02; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Malaria
Keywords: Malaria; Rapid Diagnostic Tests for Malaria; Chemical Shops; Drug Shops; Diagnostics; Testing for Malaria
MeSH Terms: conditions — Malaria | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid Diagnostic Test (Experimental): Rapid Diagnostic Test for malaria to direct antimalarial dispensing decisions in Chemical Shops
  Interventions: Procedure: Rapid Diagnostic Test
- No RDT (No Intervention): Chemical sellers dispense antimalarials as per their own decisions without the benefit of test results

INTERVENTIONS:
Procedure: Rapid Diagnostic Test — Rapid Diagnostic Test for Malaria carried out to direct antimalarial dispensing. No antimalarials for negative tests, antimalarials for positive tests
  Other Names: mRDT; RDT for malaria; RDT
  Arms: Rapid Diagnostic Test

SUMMARY:
This study aims to test directly by means of a cluster randomized controlled trial, the impact of the introduction of RDTs for malaria on dispensing behaviour of chemical sellers, the main non-formal outlet for drugs locally, at community level.

DETAILED DESCRIPTION:
In many settings the majority of people with malaria particularly the poorest do not access formal care but access anti-malarials at the informal community level. ACTs were previously unaffordable to this group but this should change with the introduction of the AMFm. To avoid missing alternative causes of illness, reduce costs and delay the spread of resistance to ACTs, they need to be targeted at those who really need them. Studies in formal healthcare settings in Ghana have shown that where microscopy is not available, the impact of Rapid Diagnostic Tests (RDTs) can be substantial. RDTs are relatively simple to use, requiring fairly minimal training to master the mechanics of test preparation and interpretation Whether to deploy RDTs as part of AMFm is unclear at this time.Even in the absence of AMFm the question about how best to target antimalarials in the community is an important one, and will get more so as malaria incidence in many countries decreases, making presumptive treatment of all febrile illness as malaria increasingly ineffective. Locally chemical sellers are the closest equivalent as they provide the majority of treatments, especially for the poorest.

It is difficult to predict whether RDTs would make chemical sellers more commonly accessed (because patients prefer a diagnosis) , or less accessed (patients do not like having choice restricted/do not want a blood test etc). Studies in other settings suggest interventions to improve diagnosis by shop-keepers can be effective and cost-effective .

ELIGIBILITY:
Inclusion Criteria:

* Patients reporting to chemical seller with complaint of fever or who request for an anti-malarial drug

Exclusion Criteria:

* Clients providing a prescription from a health facility
* Clients with signs of severe disease who will be referred onward

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4748 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The proportion of clients negative for malaria by double read research blood slide who received an anti-malarial in both arms | Until the estimated sample size is obtained or up to 2 yrs whichever comes first
  Out of all clients who test negative when their blood slides are read by two independent expert microscopists, how many received an antimalarial treatment from the Licensed Chemical Seller

SECONDARY OUTCOMES:
Proportion of mRDT -ve clients who received an anti-malarial in the RDT arm | Until the estimated sample size is obtained or up to 2 years, whichever comes first
  Out of all clients who test negative by RDT, number who receive an antimalarial
Proportion of clients tested using a Rapid Diagnostic Test | Until the estimated sample size is obtained or up to 2 years, whichever comes first
  The number of clients who agree to be tested with an RDT Out of all clients who meet inclusion criteria
Proportion of clients in each arm receiving an antibiotic | Until the estimated sample size is obtained or up to 2 years, whichever comes first
  The number of clients in the intervention and control arms who receive an antibiotic out of the total number of clients recruited into each arm
Proportion of clients receiving addittional or alternative treatments to antimalarial and which these are | Until the estimated sample size is obtained or up to 2 years, whichever comes first
  The number of clients who receive additional or alternative treatments in the intervention and control arms out of the total number recruited into both arms

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn K Ansah, MD,MPH,PhD, Principal Investigator — Ghana Health Services; Christopher C Whitty, BSc,MSc,PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Margaret Gyapong, BSc,MSc,PhD, Principal Investigator — Ghana Health Services
Locations (1):
- Dodowa Health Research Centre, Ghana Health Service, Dodowa, Greater Accra Region, Ghana

REFERENCES:
- [Derived] Ansah EK, Narh-Bana S, Affran-Bonful H, Bart-Plange C, Cundill B, Gyapong M, Whitty CJ. The impact of providing rapid diagnostic malaria tests on fever management in the private retail sector in Ghana: a cluster randomized trial. BMJ. 2015 Mar 4;350:h1019. doi: 10.1136/bmj.h1019. PMID 25739769
- See also: Malaria Capacity Development Consortium — http://www.mcdconsortium.org